CLINICAL TRIAL: NCT02343185
Title: Effects of Diaphragmatic Manual Therapy in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Eva Segura Ortí, PhD, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEU-UCH-125
Record Dates: First submitted 2014-12-22; First posted 2015-01-21 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Low Back Pain
Keywords: diaphragm; osteopathic treatment; myofascial release
MeSH Terms: conditions — Low Back Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- diaphragmatic treatment (Experimental): Subjects in this arm receive different manual techniques for the low back pain and diaphragmatic treatment.
  Interventions: Other: manual therapy with diaphragmatic treatment
- Placebo (Placebo Comparator): Subjects in this arm receive different manual techniques for the low back pain and a sham diaphragmatic treatment.
  Interventions: Other: Placebo treatment

INTERVENTIONS:
Other: manual therapy with diaphragmatic treatment — Subjects receive five sesions of manual therapy for low back pain combined with diaphragmatic treatment.
  Arms: diaphragmatic treatment
Other: Placebo treatment — Subjects receive five sesions of manual therapy for low back pain combined with a sham diaphragmatic treatment.
  Arms: Placebo

SUMMARY:
This study is a double-blind randomized clinical trial with two arms which aims to study the effects of diaphragmatic treatment in patients with nonspecific low back pain.

Low back pain has a great importance in today's society, and it is therefore important to develop an effective treatment for this condition. People with chronic nonspecific low back pain, can present respiratory disorders and get anxiety states, affecting mainly the diaphragm muscle. Therefore, given its direct anatomic relationship, the diaphragm may be part of the development of chronic low back pain. Although clinical practice guidelines for chronic low back pain have been developed, it hasn't been explored before a physiotherapy treatment especially aimed at a diaphragmatic treatment.

A double-blind randomized clinical trial with two arms will be used for this purpose, 64 patients with nonspecific low back pain referred from different hospitals of Castellón will be randomized into two groups:

* Diaphragmatic intervention with osteopathic manual therapy treatment (D).
* Diaphragmatic intervention with placebo treatment group (P).

An osteopathic manual therapy protocol for the treatment of back pain including techniques for the diaphragm muscle will be applied to the patients in group D, in a total of 5 sessions. For patients in group P, the same protocol will be performed on the diaphragm but with placebo treatment techniques.

The study focuses on the analysis of the following variables: scores on the questionnaires:

* Pain: McGill Pain Questionnaire and VAS (Visual Analogical Scale ).
* Fear Avoidance: (FABQ)
* Disability: Oswestry Disability Index and Roland-Morris
* Anxiety: HADS: (Hospital Anxiety and Depression Scale)
* Catastropizing: PCS (Pain Catastropizing Scale)
* Satisfaction with treatment (Escala de Satisfacción con el tratamiento)

The results of these pre-intervention and post-intervention variables will be compared between the two groups in the first session, in the fourth session and in the first and third month after the first intervention. The VAS score will also be assessed in the second and third session.

ELIGIBILITY:
Inclusion Criteria:

* low back pain for more than 3 months

Exclusion Criteria:

* vertebra fracture
* systemic disease
* spinal surgery
* degenerative articular disease
* acute soft tissue inflammation
* radiculopathy
* structural spine deformities
* pregnancy
* mental disease
* dermatologic disease
* rejection to manual contact

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Pain | 4 weeks
  Short form McGill Pain Questionnaire
Disability | 4 weeks
  Oswestry Disability Index

SECONDARY OUTCOMES:
Fear Avoidance Beliefs Questionnaire | 4 weeks
  FABQ
Hospital Anxiety and Depression Scale | 4 weeks
Pain Catastropizing Scale | 4 weeks
Satisfaction with treatment Questionnaire | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Juan Francisco Lisón, PhD, Study Director — University CEU UCH
Locations (1):
- University CEU UCH, Moncada, Valencia, Spain

REFERENCES:
- [Background] Assendelft WJ, Morton SC, Yu EI, Suttorp MJ, Shekelle PG. Spinal manipulative therapy for low back pain. A meta-analysis of effectiveness relative to other therapies. Ann Intern Med. 2003 Jun 3;138(11):871-81. doi: 10.7326/0003-4819-138-11-200306030-00008. PMID 12779297
- [Background] Waddell G, Newton M, Henderson I, Somerville D, Main CJ. A Fear-Avoidance Beliefs Questionnaire (FABQ) and the role of fear-avoidance beliefs in chronic low back pain and disability. Pain. 1993 Feb;52(2):157-168. doi: 10.1016/0304-3959(93)90127-B. PMID 8455963
- [Background] Herrero MJ, Blanch J, Peri JM, De Pablo J, Pintor L, Bulbena A. A validation study of the hospital anxiety and depression scale (HADS) in a Spanish population. Gen Hosp Psychiatry. 2003 Jul-Aug;25(4):277-83. doi: 10.1016/s0163-8343(03)00043-4. PMID 12850660
- [Background] Andersson GB, Lucente T, Davis AM, Kappler RE, Lipton JA, Leurgans S. A comparison of osteopathic spinal manipulation with standard care for patients with low back pain. N Engl J Med. 1999 Nov 4;341(19):1426-31. doi: 10.1056/NEJM199911043411903. PMID 10547405
- [Background] Airaksinen O, Brox JI, Cedraschi C, Hildebrandt J, Klaber-Moffett J, Kovacs F, Mannion AF, Reis S, Staal JB, Ursin H, Zanoli G; COST B13 Working Group on Guidelines for Chronic Low Back Pain. Chapter 4. European guidelines for the management of chronic nonspecific low back pain. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S192-300. doi: 10.1007/s00586-006-1072-1. No abstract available. PMID 16550448
- [Derived] Marti-Salvador M, Hidalgo-Moreno L, Domenech-Fernandez J, Lison JF, Arguisuelas MD. Osteopathic Manipulative Treatment Including Specific Diaphragm Techniques Improves Pain and Disability in Chronic Nonspecific Low Back Pain: A Randomized Trial. Arch Phys Med Rehabil. 2018 Sep;99(9):1720-1729. doi: 10.1016/j.apmr.2018.04.022. Epub 2018 May 19. PMID 29787734